

## **Informed Consent Form**

(Copy to parents or guardians)

| I, | (name of the parent or guardian), agree |
|---|---|
| with the participation of | |
| | intervention programs on preschoolers' social-emotional competence" |
| implemented by Andreia Rodrigues, Maste | er in Psychomotricity, and supervised by Professor Dr. Guida Veiga, Professo |
| Dr. José Marmeleira, and Professor Dr. Clar | inda Pomar. This study was approved by the Direction Board of the school and |
| by the Ethics Committee of the University of | of Évora. |
| The intervention programs focus | on relaxation activities and/or in loose parts play, being implemented in the |
| school. Before and after the intervention | programs some measurements will be collected to examine the impact or |
| children's' social-emotional outcomes. | |
| All instruments will be collected by | y the same researcher throughout the different stages of testing, in the school |
| In this way, filmed tasks will be applied to c | children (e.g., emotion identification through some drawings of facial emotion |
| expressions), and questionnaires will be g | given to parents or guardians and teachers to understand the effects of the |
| intervention programs on children's social- | emotional development. |
| By participating in this study, I will | l be contributing to the fulfillment of scientific research with social value, tha |
| will enable new knowledge about prescho | ool education and contribute to the promotion of children's health and well- |
| being. | |
| | uments used directly and individually with children do not interfere with their |
| | engage positively during their application. My participation and my child's |
| | vithdraw at any time, or refuse to participate with no consequences. I was |
| | nalyzed confidentially. The results of this study may be published in a scientific |
| <del>-</del> | ne child, but the group of children that participated in the study. However, if |
| <b>authorize it</b> , the images collected may be ι | use for the purpose of disseminating the study. |
| I understand the procedures. | |
| I will be able to request more informati | on about the study through the contacts of the responsible researcher |
| andreia.s.rodri@gmail.com (965388789). | on about the stady through the contacts of the responsible researcher |
| Please scratch the option that does not ma | tter: |
| I authorize / I do not authorize my child t | o participate in the study. |
| I authorize / I do not authorize the collec | ted video/images to be used for the dissemination of the study. |
| Date: 01/11/2021 | |
| Signature: | |
| Responsible researcher signature: | |
| | <del></del> |



## **Informed Consent Form**

(Copy to investigation group)

| I, (name of the parent or guardian), agree |
|---|
| with the participation of (name of the child) in the |
| study "Effects of three body-oriented intervention programs on preschoolers' social-emotional competence" |
| implemented by Andreia Rodrigues, Master in Psychomotricity, and supervised by Professor Dr. Guida Veiga, Professo |
| Dr. José Marmeleira, and Professor Dr. Clarinda Pomar. This study was approved by the Direction Board of the school and |
| by the Ethics Committee of the University of Évora. |
| The intervention programs focus on relaxation activities and/or in loose parts play, being implemented in the |
| school. Before and after the intervention programs some measurements will be collected to examine the impact or |
| children's' social-emotional outcomes. |
| All instruments will be collected by the same researcher throughout the different stages of testing, in the school |
| In this way, filmed tasks will be applied to children (e.g., emotion identification through some drawings of facial emotion |
| expressions), and questionnaires will be given to parents or guardians and teachers to understand the effects of the |
| intervention programs on children's social-emotional development. |
| By participating in this study, I will be contributing to the fulfillment of scientific research with social value, tha |
| will enable new knowledge about preschool education and contribute to the promotion of children's health and well |
| being. |
| Similar studies show that the instruments used directly and individually with children do not interfere with thei |
| well-being and that they have fun and engage positively during their application. My participation and my child' |
| participation are voluntary, and we can withdraw at any time, or refuse to participate with no consequences. I wa |
| assured that all data will be collected and analyzed confidentially. The results of this study may be published in a scientification of the collected and analyzed confidentially. |
| journal. Published data will not concern one child, but the group of children that participated in the study. However, if |
| authorize it, the images collected may be use for the purpose of disseminating the study. |
| I understand the procedures. |
| I will be able to request more information about the study through the contacts of the responsible researcher |
| andreia.s.rodri@gmail.com (965388789). |
| Please scratch the option that does not matter: |
| I authorize / I do not authorize my child to participate in the study. |
| I authorize / I do not authorize the collected video/images to be used for the dissemination of the study. |
| Date: 01/11/2021 |
| Signature: |
| Responsible researcher signature: |